CLINICAL TRIAL: NCT02591771
Title: Phase II Clinical Trial for a Stepwise Progression in the Treatment of Cardiogenic Shock
Brief Title: Study of Multistep Pharmacological and Invasive Management for Cardiogenic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Niguarda Hospital (Other)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AltShock
Record Dates: First submitted 2015-10-11; First posted 2015-10-30 (Estimated); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Cardiogenic Shock
Keywords: Adrenaline; Extra Corporeal Life Support; Inotropes
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adrenaline (Experimental): i.v. adrenaline infusion as an early and fast haemodynamic stabilizer, associated with a tight tissue perfusion monitoring, in the context of a stepwise progression in the treatment of cardiogenic shock, including ventricular mechanical support
  Interventions: Drug: adrenaline

INTERVENTIONS:
Drug: adrenaline — i.v. adrenaline infusion as an early and fast haemodynamic stabilizer, associated with a tight tissue perfusion monitoring, in the context of a stepwise progression in the treatment of cardiogenic shock, including ventricular mechanical support

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of i.v. adrenaline infusion as an early and fast haemodynamic stabilizer, associated with a tight tissue perfusion monitoring, in the context of a stepwise progression in the treatment of cardiogenic shock, including ventricular mechanical support.

DETAILED DESCRIPTION:
Cardiogenic shock is characterized by a decrease in cardiac output and increased ventricular pressures, with subsequent symptoms and signs of systemic hypoperfusion. In spite of the multiple pharmacological chances the in-hospital mortality rate is still very high (around 60% of patients) and nowadays there is not a therapeutic "reference standard" associated with an improved survival at short and midterm. Adrenaline is a mainstay of resuscitation therapy during cardiopulmonary arrest, however, it is not clear whether this inotrope actually facilitates an improvement in patients affected by cardiogenic shock. In a small local evidence-based experience, contrary to current opinion, it has been shown that adrenaline may still have a role in the treatment of patients with low output state. This phase II study tests the hypothesis that adrenaline infusion, integrated in a multistep approach at increasing intensity, can be a valid support with limited side effects.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 and < 75, men and women;
* 1) SBP < 90mmHg or MAP < 60 mmHg, after an appropriate fluid challenge if there is no sign of overt fluid overload; OR 2) need of vasoactive agents to maintain SBP > 90 mmHg or MAP > 60 mmHg.
* Pre-existing diagnosis of heart failure with reduced ejection fraction (left ventricle systolic function ≤35%).
* Moreover, eligible patients have to fit at least ONE of the following criteria/items of overt hypoperfusion: mixed venous oxygen saturation < 60%; arterial lactates > 2 mmol/L; oliguria < 0.5 ml/Kg/h for at least 6 hours.
* Eligible patients shouldn't have contraindications to HRT.

Exclusion Criteria

* Cardiogenic shock symptoms beyond 6 hours.
* Septic shock with evident septic focus.
* Cardiogenic shock due to acute myocardial infarction.
* Cardiogenic shock due to acute myocarditis.
* Cardiogenic shock due to pulmonary thromboembolism.
* Reiterating major arrhythmias: VT or VF or AF, with ventricular rate > 160 bpm.
* Severe aortic valve disease.
* Obstructive hypertrophic cardiomyopathy or constrictive pericarditis or severe heart failure due to congenital heart disease
* Severe peripheral vascular disease that contraindicates mechanical support insertion.
* Cardiogenic shock secondary to either cardiac or non-cardiac surgery.
* Post-cardiac arrest syndrome following out of hospital cardiac arrest
* Comorbidities with ominous prognosis (life expectancy < 1 year).
* End-stage organ failure.
* Pregnant, lactating or subjects planning pregnancy during the course of the trial.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Survival at 60 days | 60 days
  number of successes

SECONDARY OUTCOMES:
Duration of i.v. infusion with adrenaline | 30 days
Adrenaline maximum dose | 30 days
Time to weaning from beginning with pharmacological therapy and mechanical ventricular support | 30 days
Length of stay | 30 days
Sum of medical staff support and nursing-care hours dedicated to each patient | Within patient hospitalization, each day from day 1 to day 30
Membrane oxygenation | 60 days
  Escalation to venoarterial extracorporeal membrane oxygenation (VA-ECMO)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Niguarda Hospital, Milan, MI
  - Ospedale San Raffaele, Milan

REFERENCES:
- [Result] Morici N, Oliva F, Ajello S, Stucchi M, Sacco A, Cipriani MG, De Bonis M, Garascia A, Gagliardone MP, Melisurgo G, Russo CF, La Vecchia C, Frigerio M, Pappalardo F. Management of cardiogenic shock in acute decompensated chronic heart failure: The ALTSHOCK phase II clinical trial. Am Heart J. 2018 Oct;204:196-201. doi: 10.1016/j.ahj.2018.07.009. Epub 2018 Jul 20. PMID 30100052